CLINICAL TRIAL: NCT03822598
Title: Implementation and Evaluation of Teaching Recovery Techniques (TRT) Among Asylum-seeking and Refugee Children
Brief Title: Promoting Asylum-seeking and Refugee Children's Coping With Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: University of Tromso (Other); University of Bergen (Other); Norwegian Directorate of Children, Youth, and Family Affairs (Unknown); Norwegian Directorate of Immigration (Unknown); Norwegian Directorate of Integration and Diversity (Unknown)
Responsible Party: Principal Investigator, Brit Oppedal, Principal Investigator, Norwegian Institute of Public Health
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 16/54571
Record Dates: First submitted 2019-01-21; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Mental Health Disorder; Post-Traumatic Stress Disorder in Adolescence; Depression; Social Anxiety
Keywords: Teaching Recovery Techniques; Asylum-seeking children; Refugee children; Low-threshold intervention
MeSH Terms: conditions — Mental Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Two stages of recruitment: 1) We recruited asylum reception centers and refugee resettlement municipalities located all over Norway 2) Invite asylum-seeking and refugee children in these institutions to participate, and assigning them by intstitution to control and intervention conditions. The intervention groups started implementing TRT between late September and late October. The control groups started implementing TRT between medio November and beginning of February.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Teaching Recovery Techniques implemented 1- 3 weeks after recruitment
  Interventions: Behavioral: Teaching Recovery Techniques, TRT
- Wait-list control group (Active Comparator): Delayed implementation of Teaching Recovery Techniques (after the experimental group has completed the program)
  Interventions: Behavioral: Teaching Recovery Techniques, TRT

INTERVENTIONS:
Behavioral: Teaching Recovery Techniques, TRT — TRT is a , low-threshold, group based, manual driven short term intervention to reduce trauma-related mental health problems. The program is based on principles from trauma-focused cognitive-behavioral therapy

SUMMARY:
A short term trauma-focused cognitive- behavioral program to reduce trauma-related mental health problems among asylum-seeking and refugee children.

The main hypothesis of the study is that the TRT program significantly improves mental health (i.e. reduces symptoms of post-traumatic symptoms, depression and generalized anxiety and increases perceived quality of life (Qol) in the intervention group compared to the waiting-list control group.

DETAILED DESCRIPTION:
Teaching Recovery Techniques (TRT) was developed by Children and War Foundation (www.childrenandwarfoundation.org ) as a tool to support children in coping with their mental reactions to being exposed to war and catastrophes. TRT has proven to be effective in reducing trauma-related mental health symptoms in such contexts. However, it has never been used with children experiencing all the uncertainties and stress of an asylum-seeking context, or with refugee children in high-income countries. The main aim of the present study is therefore to implement and evaluate the TRT among asylum-seeking and refugee children in the context of four different care conditions: 1)asylum-seeking children who arrived accompanied by a legal care-taker 2) asylum-seeking children less than 15 years in care centers administered by the Child Welfare Services 3) asylum-seeking children 15 years and older living in asylum centers regulated by the Directorate of Immigration 4) Former unaccompanied asylum-seeking children who have been granted residence (refugees) and are resettled in a municipality in Norway.

Based on Power analyses, the target group is 40 children in each care condition (total n = 160) > 9 years speaking Arabic, Tigrinya, Somali, Dari, or Pashto.

The study employs a randomized clustered experimental design that includes a waiting list control group, which will receive the TRT when the intervention group has completed the program.

ELIGIBILITY:
Inclusion Criteria:

* Accompanied asylum-seeking children living in reception centers,
* Unaccompanied asylum-seeking children living in reception centers
* Unaccompanied refugee minors who have been granted residence

Children in the target Groups reported symptoms of post-traumatic stress above clinical cut-off on Children's Revised Impact of Event Scale, 8 items

-

Exclusion Criteria:

* Psychosis,
* Mental disabilities

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Children's Revised Impact of Event Scale (CRIES-13) | Change in CRIES-13 scores from baseline (T1) to two weeks (T2) and two months after intervention is completed.
  Self-reported symptoms of intrusion, hyperarousal and avoidance. ' The participants check how often during the last week they had each symptom from "never" (0); "rarely" (1) "sometimes" (3) and "frequently" (5)

SECONDARY OUTCOMES:
Screen for Child Anxiety Related Disorders (SCARED). 9 items tapping symptoms of generalized anxiety disorder, and 7 items tapping symptoms of social anxiety | Change in SCARED-scores from baseline (T1) to two weeks (T2) and two months after intervention is completed.
  Measures if children have perceived each anxiety symptom over the last three months from "not true, or hardly ever true" (0), "somewhat true or sometimes true" (1) "very true or often true" (2)
Cantril Ladder | Change in scores from baseline (T1) to two weeks (T2) and two months after intervention is completed.
  Measures current subjective well-being on a ladder With 11 steps from "worst possible life" (0) to "best possible life" (10)
Montgomery-Aasberg Depression Scale, MADRS | Change in MADRS-scores from baseline (T1) to two weeks (T2) and two months after intervention is completed.
  9 items assessing patients' mood, feelings of unease, sleep, appetite, ability to concentrate, initiative, emotional involvement, pessimism and zest for life over the last three days. Each item is scored between 0 (not a problem for me) and 3 (affects me very much), with three intermediate levels (0.5, 1.5, 2.5).

CONTACTS AND LOCATIONS:
Locations (16):
- Norway (16):
  - Bergen Municipality, Bergen
  - Nordre Land municipality, Dokka
  - Drammen Municipality, Drammen
  - Engerdal Municipality, Drevsjø
  - Fredrikstad municipality, Fredrikstad
  - Gjøvik municipality, Gjøvik
  - Ringerike Municipality, Hønefoss
  - Grue municipality, Kirkenær
  - Levanger municipality, Leira
  - Lyngdal municipality, Lyng
  - Lyngdal municipality, Lyngdal
  - Bærum municipality, Rud
  - Salten municipality, Sjøvegan
  - Stavanger municipality, Stavanger
  - Trondheim municipality, Trondheim
  - Vadsø municipality, Vadsø

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make Individual Patient Data (IPD) available. If IPD are to be shared, we follow the regulations of the Norwegian Institute of Public Health

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03822598/Prot_SAP_000.pdf